CLINICAL TRIAL: NCT06407778
Title: Comparison of Effects of High Intensity Strength Training and Muscle Energy Technique on Pain, ROM and Functional Status in Patients With Total Knee Replacement
Brief Title: Comparison of High Intensity Strength Training and Muscle Energy Techniques in TKR Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01104
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis; Arthroplasty, Knee Replacement; Resistance Training
Keywords: Total Knee Replacement; Knee Osteoarthritis; Strength Training; Muscle Energy Technique
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome Assessor will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Strength Training (Experimental): Group of TKR patients are given high intensity strength training.
  Interventions: Other: High Intensity Strength Training
- Muscle Energy Technique Exercises (Active Comparator): patients are given muscle energy technique exercise.
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: High Intensity Strength Training — * High-intensity workouts to strengthen the quadriceps and enhance knee function;
  * Knee flexion and extension 10 lbs.
  * 10RM of hip flexion and extension
  * 10RM hip adduction and abduction
  * Standing with feet aligned for one minute*2, standing on one leg's forefoot and the other leg's heel for two minutes*2, standing on one foot for three seconds*15, and walking ten meters in a straight line for four minutes
  * 4-week program; 3 days/week; Conventional Treatment: Exercises for range of motion, mobility and weight bearing, muscle stretching, static quadriceps exercise, quadriceps exercise, and straight leg raising
  Arms: High Intensity Strength Training
Other: Muscle Energy Technique — The Muscle Energy Technique (MET) to strengthen and flex your quadriceps and hamstrings.
  * After maintaining an isometric contraction for ten seconds, a little stretch was maintained for thirty seconds.
  * Four contractions every treatment, separated by three seconds of rest. Standing with feet parallel for one minute*2, standing on one leg's forefoot and the other leg's heel for two seconds*2, standing on the forefoot for three seconds*15
  * Move in a 10 m by 4 straight line.
  * 4-week program; 3 days/week Conventional Treatment: Exercises for range of motion, mobility and weight bearing, muscle stretching, static quadriceps exercise, quadriceps exercise, and straight leg raising
  Arms: Muscle Energy Technique Exercises

SUMMARY:
Globally, the prevalence of total joint replacement (TKR) procedures has been rising, providing patients with better joint function, decreased pain, and enhanced quality of life. A thorough and successful postoperative rehabilitation program, which attempts to restore optimal function and lower the risk of problems related to the treatment, is necessary for the success of total knee replacement (TKR) procedures. After total knee replacement, postoperative rehabilitation is a crucial stage in the patient's healing process. Normal knee function is frequently hampered by issues like pain management, muscular weakness, joint stiffness, and proprioceptive deficiencies. Therefore, choosing a suitable rehabilitation regimen is crucial.

DETAILED DESCRIPTION:
The main objective of this study is to compare two different rehabilitation strategies: Muscle Energy Techniques with Balance Exercises and High Intensity Strength Training with Balance Exercises. The research aims to maximize postoperative results for patients who have undergone total knee replacement surgery.

The focus on resistance exercises intended to improve muscle strength and power is what defines high intensity strength training, or HIST. Research has indicated that HIST is beneficial in enhancing joint stability, muscle function, and overall functional outcomes across a range of orthopedic groups. Its precise use and effect on patients recovering from TKR surgery, however, need further investigation. In order to increase joint mobility, lessen pain, and improve neuromuscular control, patients who get Muscle Energy Techniques (MET) actively participate in targeted muscle contractions. MET has demonstrated potential in treating muscular imbalances.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 45 and 75
* Patients should be within a certain timeframe following surgery (e.g., post op day 0-day) to ensure homogeneity throughout the rehabilitation phase.
* Patients who have had primary total knee replacement
* To take part in the RCT, participants must give informed consent
* they must be able and willing to follow the study protocol's instructions for post-rehabilitation care.

Exclusion Criteria:

* Comorbidities: Individuals with significant comorbidities affecting rehabilitation, such as severe cardiovascular disease or neuromuscular disorders, may be excluded.
* Allergies/Contraindications: Patients with allergies or contraindications to specific exercises or techniques used in the study.
* Inadequate Cognitive Function: Participants with cognitive impairments that prevent them from comprehending and adhering to the rehabilitation protocols.
* Other Knee Surgeries: Patients who have had other knee surgeries or have had bilateral knee replacements may be excluded due to variations in recovery and rehabilitation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
ROM | 4th week
  An instrument called a goniometer will be used to measure angles or rotate objects into desired positions. In orthopedics, it is primarily used to quantify joint angles.
  Changes from the baseline was taken.
Functional Status: Knee Injury and Osteoarthritis outcome score | 4th week
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic scales, and generic measures. Scores between 0 and 100 represent the percentage of the total possible score achieved.
Pain : Numeric Pain Rating Scale | 4th week
  A simple tool for measuring pain intensity is the Numeric Pain Rating Scale. This grading system has eleven points: zero represents no pain, and ten represents the "worst pain imaginable or highest level of discomfort.
  Changes from the baseline was taken.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Amna Tariq, DPT, Principal Investigator — Riphah International University
Locations (1):
- Horizon Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun JN, Shan YZ, Wu LX, Li N, Xu FH, Kong XR, Zhang B. Preoperative high-intensity strength training combined with balance training can improve early outcomes after total knee arthroplasty. J Orthop Surg Res. 2023 Sep 15;18(1):692. doi: 10.1186/s13018-023-04197-3. PMID 37715204
- [Background] Casana J, Calatayud J, Ezzatvar Y, Vinstrup J, Benitez J, Andersen LL. Preoperative high-intensity strength training improves postural control after TKA: randomized-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1057-1066. doi: 10.1007/s00167-018-5246-2. Epub 2018 Oct 25. PMID 30361758
- [Background] Irrgang JJ, Snyder-Mackler L, Wainner RS, Fu FH, Harner CD. Development of a patient-reported measure of function of the knee. J Bone Joint Surg Am. 1998 Aug;80(8):1132-45. doi: 10.2106/00004623-199808000-00006. PMID 9730122
- [Background] Bade MJ, Stevens-Lapsley JE. Early high-intensity rehabilitation following total knee arthroplasty improves outcomes. J Orthop Sports Phys Ther. 2011 Dec;41(12):932-41. doi: 10.2519/jospt.2011.3734. Epub 2011 Sep 30. PMID 21979411